CLINICAL TRIAL: NCT00415636
Title: A Phase 1 Dose-Escalation Study to Examine the Safety and Tolerability of IC83/LY2603618 Administered After Pemetrexed 500 mg/m2 Every 21 Days in Patients With Cancer
Brief Title: Safety and Tolerability of IC83/LY2603618 Administered After Pemetrexed 500 mg/m2 Every 21 Days in Patients With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11911; I2I-MC-JMMB (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-12-21; First posted 2006-12-25 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- LY2603618 40 mg/m^2 (4.5-hour infusion) (Experimental): LY2603618 40 milligrams per square meter (mg/m^2) was administered over the duration of 4.5 hours (30-minute bolus followed by a 4-hour infusion). Dose modifications were not allowed.
  Interventions: Drug: IC83/LY2603618; Drug: pemetrexed
- LY2603618 40 mg/m^2 (1-hour infusion) (Experimental): Based on pharmacokinetic (PK) data from Cohort 1 (LY2603618 40 mg/m^2 [4.5-hour infusion]), the LY2603618 40 mg/m^2 dose in Cohort 2 (LY2603618 40 mg/m^2 [1-hour infusion]) was repeated, but the dose was administered over the duration of 1 hour. Dose modifications were not allowed.
  Interventions: Drug: IC83/LY2603618; Drug: pemetrexed
- LY2603618 70 mg/m^2 (Experimental): Beginning with Cohort 3 (LY2603618 70 mg/m^2), dose modifications were allowed. LY2603618 70 mg/m^2 was administered over the course of 1 hour.
  Interventions: Drug: IC83/LY2603618; Drug: pemetrexed
- LY2603618 105 mg/m^2 (Experimental): Cohort 4: LY2603618 105 mg/m^2 administered over the duration of 1 hour.
  Interventions: Drug: IC83/LY2603618; Drug: pemetrexed
- LY2603618 150 mg/m^2 (Experimental): Cohort 5: LY2603618 150 mg/m^2 administered over the duration of 1 hour.
  Interventions: Drug: IC83/LY2603618; Drug: pemetrexed
- LY2603618 195 mg/m^2 (Experimental): Cohort 6: LY2603618 195 mg/m^2 administered over the duration of 1 hour.
  Interventions: Drug: IC83/LY2603618; Drug: pemetrexed

INTERVENTIONS:
Drug: IC83/LY2603618 — 40 mg/m^2 Day 1 and Day 9 of Cycle 1, Day 2 of subsequent cycles, unlimited 21-day cycles. Dose finding study: dose is escalated after a minimum of 6 participants receive 40 mg/m^2.
  Arms: LY2603618 40 mg/m^2 (1-hour infusion); LY2603618 40 mg/m^2 (4.5-hour infusion)
Drug: IC83/LY2603618 — 70 mg/m^2 Day 1 and Day 9 of Cycle 1, Day 2 of subsequent cycles, unlimited 21-day cycles.
  Arms: LY2603618 70 mg/m^2
Drug: IC83/LY2603618 — 105 mg/m^2 Day 1 and Day 9 of Cycle 1, Day 2 of subsequent cycles, unlimited 21-day cycles.
  Arms: LY2603618 105 mg/m^2
Drug: IC83/LY2603618 — 150 mg/m^2 Day 1 and Day 9 of Cycle 1, Day 2 of subsequent cycles, unlimited 21-day cycles.
  Arms: LY2603618 150 mg/m^2
Drug: IC83/LY2603618 — 195 mg/m^2 Day 1 and Day 9 of Cycle 1, Day 2 of subsequent cycles, unlimited 21-day cycles.
  Arms: LY2603618 195 mg/m^2
Drug: pemetrexed — pemetrexed 500 mg/m^2, intravenous (IV), Day 8 of Cycle 1, Day 1 of subsequent cycles, unlimited 21-day cycles
  Other Names: Alimta; LY231514
  Arms: LY2603618 40 mg/m^2 (4.5-hour infusion)
Drug: pemetrexed — pemetrexed 500 mg/m^2 IV, Day 8 of Cycle 1, Day 1 of subsequent cycles, unlimited 21-day cycles
  Arms: LY2603618 105 mg/m^2; LY2603618 150 mg/m^2; LY2603618 195 mg/m^2; LY2603618 40 mg/m^2 (1-hour infusion); LY2603618 70 mg/m^2

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of IC83/LY2603618 for the treatment of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Has at least one lesion that can be evaluated by Response Evaluation Criteria In Solid Tumors (RECIST)
* Has fully recovered from all toxicities due to the following:

  1. Local radiation therapy that ended at least 14 days prior to Cycle 1, Day 1.
  2. Surgery.
* Has a life expectancy of at least 3 months.
* Negative serum pregnancy test.

Exclusion Criteria:

* Is pregnant or breastfeeding.
* Is a woman of childbearing potential unwilling to use an approved, effective means of contraception according to the institution's standards.
* Is a man of childbearing potential unwilling to use an approved, effective means of contraception according to the institution's standards.
* Has a history of brain metastases, unless adequately treated and without radiologic evidence of progressive disease for at least 3 months after completion of therapy.
* Has a known active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-01; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM-5PM Eastern time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2603618 40 mg/m^2 (1-hour Infusion): Based on pharmacokinetic (PK) data from Cohort 1 (LY2603618 40 mg/m^2 [4.5-hour infusion]), LY2603618 40 mg/m^2 dose in Cohort 2 (LY2603618 40 mg/m^2 [1-hour infusion]) was repeated, but the dose was administered over the duration of 1 hour. Dose modifications were not allowed.
- LY2603618 105 mg/m^2: LY2603618 105 mg/m^2 administered over the duration of 1 hour.
- LY2603618 150 mg/m^2: LY2603618 150 mg/m^2 administered over the duration of 1 hour.
- LY2603618 195 mg/m^2: LY2603618 195 mg/m^2 administered over the duration of 1 hour.
Period: Overall Study
Arm/Group | LY2603618 40 mg/m^2 (4.5-hour Infusion) | LY2603618 40 mg/m^2 (1-hour Infusion) | LY2603618 70 mg/m^2 | LY2603618 105 mg/m^2 | LY2603618 150 mg/m^2 | LY2603618 195 mg/m^2
Started | 3 | 3 | 3 | 13 | 6 | 3
Completed | 2 (Completed = Participant received 2 cycles of treatment) | 3 (Completed = Participant received 2 cycles of treatment) | 2 (Completed = Participant received 2 cycles of treatment) | 7 (Completed = Participant received 2 cycles of treatment) | 4 (Completed = Participant received 2 cycles of treatment) | 1 (Completed = Participant received 2 cycles of treatment)
Not Completed | 1 | 0 | 1 | 6 | 2 | 2
Not completed — Symptomatic deterioration | 1 | 0 | 1 | 2 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Disease progression | 0 | 0 | 0 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2603618 40 mg/m^2 (4.5-hour Infusion) | LY2603618 40 mg/m^2 (1-hour Infusion) | LY2603618 70 mg/m^2 | LY2603618 105 mg/m^2 | LY2603618 150 mg/m^2 | LY2603618 195 mg/m^2 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 13 | 6 | 3 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (6.24) | 58.0 (10.54) | 48.3 (16.07) | 60.6 (9.95) | 63.5 (11.04) | 55.7 (18.77) | 58.1 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 5 | 3 | 1 | 15
  Male | 0 | 2 | 1 | 8 | 3 | 2 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 3 | 12 | 6 | 3 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 2 | 3 | 2 | 13 | 6 | 2 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 3 | 13 | 6 | 3 | 31
Primary Cancer Type [Count of Participants; unit: Participants]
  Breast | 3 | 1 | 1 | 0 | 1 | 0 | 6
  Non-small Cell Lung | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Pancreatic | 0 | 0 | 0 | 3 | 2 | 1 | 6
  Other | 0 | 2 | 2 | 9 | 3 | 2 | 18
Eastern Cooperative Oncology Group (ECOG) Rating at Screening [Count of Participants; unit: Participants] — Classifies participants according to their functional impairment. Scores range from 0 to 5: 0=Fully Active; 1=Ambulatory, Restricted Strenuous Activity; 2=Ambulatory, No Work Activities; 3=Partially Confined to Bed, Limited Self Care; 4=Completely Disabled; 5=Death.
  Participants
    ECOG Rating 0 | 2 | 1 | 0 | 4 | 1 | 0 | 8
    ECOG Rating 1 | 1 | 2 | 3 | 9 | 5 | 3 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Summary tables of serious AEs (SAEs) and all other non-serious adverse events (AEs) are located in the Reported Adverse Event Module.
Time Frame: baseline up to 24 months
Population: The safety population was comprised of all participants who received any amount of LY2603618.
Measure: Count of Participants; unit: Participants
Groups:
- LY2603618 40 mg/m^2 (4.5-hour Infusion): 4.5-hour intravenous (IV) infusion of IC83/LY2603618 40 mg/m^2
- LY2603618 40 mg/m^2 (1-hour Infusion): 1.0-hour IV infusion of IC83/LY2603618 40 mg/m^2
- LY2603618 70 mg/m^2: 1.0-hour IV infusion of IC83/LY2603618 70 mg/m^2
- LY2603618 105 mg/m^2: 1.0-hour IV infusion of IC83/LY2603618 105 mg/m^2
- LY2603618 150 mg/m^2: 1.0-hour IV infusion of IC83/LY2603618 150 mg/m^2
- LY2603618 195 mg/m^2: 1.0-hour IV infusion of IC83/LY2603618 195 mg/m^2
Arm/Group | LY2603618 40 mg/m^2 (4.5-hour Infusion) | LY2603618 40 mg/m^2 (1-hour Infusion) | LY2603618 70 mg/m^2 | LY2603618 105 mg/m^2 | LY2603618 150 mg/m^2 | LY2603618 195 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 13 | 6 | 3
Participants
  Other Non-Serious Adverse Events (AEs) | 3 | 3 | 3 | 13 | 6 | 3
  Serious Adverse Events (SAEs) | 1 | 0 | 2 | 8 | 4 | 2

2. Secondary Outcome: Pharmacokinetic (PK) Parameter: Maximum Observed Plasma Concentration (Cmax) of IC83/LY2603618
Description: Cmax was estimated from the plasma concentration data of LY2603618 versus time profiles.
Time Frame: Day 1 and Day 9 of Cycle 1
Population: Pharmacokinetic (PK) analyses were conducted for individual participants who received at least 1 dose of study drug and had PK samples collected.
Measure: Mean (Standard Deviation); unit: nanograms per millimeter (ng/mL)
Groups:
- LY2603618 40 mg/m^2 (4.5-hour Infusion): 4.5-hour intravenous (IV) infusion of IC83/LY2603618 40 mg/m^2 on Day 1 (alone) and Day 9 of Cycle 1.
- LY2603618 40 mg/m^2 (1-hour Infusion): 1.0-hour IV infusion of IC83/LY2603618 40 mg/m^2 on Day 1 (alone) and Day 9 of Cycle 1.
- LY2603618 70 mg/m^2: 1.0-hour IV infusion of IC83/LY2603618 70 mg/m^2 on Day 1 (alone) and Day 9 of Cycle 1.
- LY2603618 105 mg/m^2: 1.0-hour IV infusion of IC83/LY2603618 105 mg/m^2 on Day 1 (alone) and Day 9 of Cycle 1.
- LY2603618 150 mg/m^2: 1.0-hour IV infusion of IC83/LY2603618 150 mg/m^2 on Day 1 (alone) and Day 9 of Cycle 1.
- LY2603618 195 mg/m^2: 1.0-hour IV infusion of IC83/LY2603618 195 mg/m^2 on Day 1 (alone) and Day 9 of Cycle 1.
Arm/Group | LY2603618 40 mg/m^2 (4.5-hour Infusion) | LY2603618 40 mg/m^2 (1-hour Infusion) | LY2603618 70 mg/m^2 | LY2603618 105 mg/m^2 | LY2603618 150 mg/m^2 | LY2603618 195 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 13 | 6 | 3
nanograms per millimeter (ng/mL)
  Day 1 | 578 (181) | 1560 (358) | 2310 (1330) | 4220 (1370) | 4230 (1370) | 6840 (839)
  Day 9: number analyzed (Participants) | 3 | 3 | 3 | 12 | 5 | 3
  Day 9 | 614 (169) | 2010 (581) | 2510 (942) | 4540 (2270) | 3560 (1320) | 7580 (1260)

3. Secondary Outcome: Pharmacokinetic (PK) Parameter: Area Under the IC83/LY2603618 Plasma Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-∞])
Description: AUC[0-∞] was calculated from the plasma concentration data of LY2603618 versus time profiles.
Time Frame: Day 1 and Day 9 of Cycle 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | LY2603618 40 mg/m^2 (4.5-hour Infusion) | LY2603618 40 mg/m^2 (1-hour Infusion) | LY2603618 70 mg/m^2 | LY2603618 105 mg/m^2 | LY2603618 150 mg/m^2 | LY2603618 195 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 13 | 6 | 3
nanograms*hour per milliliter (ng*h/mL)
  Day 1 | 7580 (790) | 10300 (2810) | 9510 (5560) | 76400 (65000) | 61900 (53300) | 122000 (42000)
  Day 9: number analyzed (Participants) | 3 | 3 | 3 | 12 | 5 | 3
  Day 9 | 7540 (1790) | 11000 (2550) | 10900 (6280) | 52000 (33900) | 55000 (45000) | 119000 (30300)

4. Secondary Outcome: Percentage of Participants With Best Overall Response
Description: Percentage of participants with tumor response (best confirmed overall response) assessed as complete response (CR) or partial response (PR) to treatment according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria. CR=disappearance of all target lesions; PR=30% decrease in sum of longest diameter of target lesions; Progressive Disease (PD)=20% increase in sum of longest diameter of target lesions; Stable Disease (SD) =small changes that do not meet above criteria. Best Overall Response (%)=number of participants with CR+PR/number of participants in treatment arm * 100.
Time Frame: baseline up to 24 months
Population: A modified intent-to-treat population (mITT) was used to summarize the data for tumor response. The mITT population consisted of all participants who received any dose of study drug and had at least 1 nonmissing postbaseline tumor response assessment.
Measure: Number; unit: Percentage of participants
Groups:
- LY2603618 40 mg/m^2 (4.5 Hours): 4.5-hour IV infusion of IC83/LY2603618 40 mg/m^2
- LY2603618 40 mg/m^2 (1 Hour): 1.0-hour IV infusion of IC83/LY2603618 40 mg/m^2
Arm/Group | LY2603618 40 mg/m^2 (4.5 Hours) | LY2603618 40 mg/m^2 (1 Hour) | LY2603618 70 mg/m^2 | LY2603618 105 mg/m^2 | LY2603618 150 mg/m^2 | LY2603618 195 mg/m^2
Number analyzed (Participants) | 2 | 3 | 2 | 10 | 4 | 2
Percentage of participants
  Complete Response (CR) | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 0 | 10 | 0 | 0
  Stable Disease (SD) | 0 | 66.7 | 50 | 20 | 75 | 50
  Progressive Disease (PD) | 100 | 33.3 | 50 | 70 | 25 | 50
  Not Determined | 0 | 0 | 0 | 0 | 0 | 0
  Best Overall Response (CR + PR) | 0 | 0 | 0 | 10 | 0 | 0

ADVERSE EVENTS:
Arm/Group | LY2603618 40 mg/m^2 (4.5-hour Infusion) | LY2603618 40 mg/m^2 (1-hour Infusion) | LY2603618 70 mg/m^2 | LY2603618 105 mg/m^2 | LY2603618 150 mg/m^2 | LY2603618 195 mg/m^2
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 2/3 | 8/13 | 4/6 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 13/13 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2603618 40 mg/m^2 (4.5-hour Infusion) (N=3) | LY2603618 40 mg/m^2 (1-hour Infusion) (N=3) | LY2603618 70 mg/m^2 (N=3) | LY2603618 105 mg/m^2 (N=13) | LY2603618 150 mg/m^2 (N=6) | LY2603618 195 mg/m^2 (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2603618 40 mg/m^2 (4.5-hour Infusion) (N=3) | LY2603618 40 mg/m^2 (1-hour Infusion) (N=3) | LY2603618 70 mg/m^2 (N=3) | LY2603618 105 mg/m^2 (N=13) | LY2603618 150 mg/m^2 (N=6) | LY2603618 195 mg/m^2 (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (4) | 1 (1) | 3 (5) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 5 (6) | 3 (3) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 2 (2) | 2 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival pallor (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 4 (6) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 2 (3) | 1 (1) | 2 (2) | 2 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (2) | 5 (7) | 3 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (2) | 3 (6) | 7 (12) | 2 (3) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (5) | 5 (6) | 3 (4) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Fatigue (General disorders) | 0 (0) | 3 (5) | 3 (3) | 4 (5) | 5 (8) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 4 (5) | 2 (3) | 0 (0)
Tenderness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breath sounds abnormal (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node palpable (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (5) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 3 (3) | 2 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penile swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 3 (3) | 1 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campbell de morgan spots (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days